CLINICAL TRIAL: NCT01302262
Title: Does the Insula Control Smoking-induced Dopamine Release? A TMS/[11C]-PHNO Study in Humans. Part I: Smoking-induced Dopamine Release: a [11C]-(+)-PHNO PET Study in Humans.
Brief Title: Smoking-induced Dopamine Release: a [11C]-(+)-PHNO PET Study in Humans
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Bernard Le Foll, MD, PhD, CCFP, Centre for Addiction and Mental Health
Other Study IDs: 143/2010
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking-induced dopamine release; [11C]-(+)-PHNO PET Study
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (15mL)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy smokers: Healthy male and female smokers. Each subject will undergo PET scan (along with craving and anxiety questionnaires) on two conditions - Smoking and Non-smoking - on two separate visits.

SUMMARY:
This study will evaluate effects of smoking on the dopaminergic system by using PET tomography with new radioligand, [11C]-(+)-PHNO. Our primary hypothesis is that smoking a cigarette will produce dopamine release and this release can be measured using PET imaging and the [11C]-(+)-PHNO radiotracer. The secondary hypothesis is that this smoking induced dopamine release will be correlated with subjective craving and anxiety ratings.

DETAILED DESCRIPTION:
This will be a within-subjects study in healthy male and female smokers. There will be one within factor condition: Smoking and Non Smoking. Therefore, there will be a repeated measure of PET scans using [11C]-(+)-PHNO under two different conditions. Ten subjects (n=5 male and n=5 female) included in the study will come on two different days and will have a Smoking or Non smoking session performed just before the PET study. Subjective assessments will be conducted at each experimental condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females
* Regular smoking of at least 10 cigarettes, excluding ultra-low nicotine cigarettes, per day for at least two years
* Score on the Fagerstrom Test for Nicotine Dependence of 4 or more
* No intention to quit or reduce tobacco use, and no treatment for tobacco dependence currently
* No history of abuse of or dependence on any other drug, defined by DSM-IV criteria

Exclusion Criteria:

* Pregnancy
* Presence of metal objects in the body or implanted electronic devices, that preclude safe MR scanning
* Claustrophobia
* Cardiovascular or cerebrovascular diseases
* Major psychiatric disorders including mood, anxiety or psychotic disorders
* History of or current neurological illnesses including seizure disorders, migraine, multiple sclerosis, movement disorders, head trauma, CVA or CNS tumor
* Gross structural brain abnormalities as revealed by T1 weighted images
* Current use or use during the previous month of medication that may affect the CNS (e.g. neuroleptics, bupropion)
* Learning disability, amnesia or other conditions that impede memory and attention

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy smokers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
[11C]-(+)-PHNO binding potential | Up to 14 days between PET scans
  The process of imaging requires the injection of a positron-emitting radiotracer (here, [11C]-(+)-PHNO) that binds to the protein of interest (here, dopamine receptor DRD2/3) followed by the measurement of this binding using the PET scanner. Dopamine release increases DRD 2/3 occcupancy which results in decreased radiotracer's binding potential, and vice versa. [11C]-(+)-PHNO binding potential will be measured on two different conditions (Smoking vs. Non-smoking) on two separate days.

SECONDARY OUTCOMES:
Subjective reports of craving | Up to 14 days between PET scans
  Levels of subjective craving will be assessed prior to and after each condition (Smoking vs. Non-smoking) on two separate days. Minnesota Nicotine Withdrawal Scale, Tiffany Questionnaire of Smoking Urges, The Urge to Smoke scale, Tobacco Craving Questionnaire, and 21-item Visual Analogue Scale will be used.
Subjective reports of anxiety | Up to 14 days between PET scans
  Subjective reports of anxiety will be collected prior to and after each condition (Smoking vs. Non-smoking) on two separate days. State anxiety questions from the Spielberg State-Trait Anxiety Inventory will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health - 33 Russell St, Toronto, Ontario, Canada

REFERENCES:
- [Background] Brody AL, Olmstead RE, London ED, Farahi J, Meyer JH, Grossman P, Lee GS, Huang J, Hahn EL, Mandelkern MA. Smoking-induced ventral striatum dopamine release. Am J Psychiatry. 2004 Jul;161(7):1211-8. doi: 10.1176/appi.ajp.161.7.1211. PMID 15229053
- [Background] Wilson AA, McCormick P, Kapur S, Willeit M, Garcia A, Hussey D, Houle S, Seeman P, Ginovart N. Radiosynthesis and evaluation of [11C]-(+)-4-propyl-3,4,4a,5,6,10b-hexahydro-2H-naphtho[1,2-b][1,4]oxazin-9-ol as a potential radiotracer for in vivo imaging of the dopamine D2 high-affinity state with positron emission tomography. J Med Chem. 2005 Jun 16;48(12):4153-60. doi: 10.1021/jm050155n. PMID 15943487
- [Background] Le Foll B, Goldberg SR, Sokoloff P. The dopamine D3 receptor and drug dependence: effects on reward or beyond? Neuropharmacology. 2005 Sep;49(4):525-41. doi: 10.1016/j.neuropharm.2005.04.022. PMID 15963538
- [Background] Le Foll B, Schwartz JC, Sokoloff P. Dopamine D3 receptor agents as potential new medications for drug addiction. Eur Psychiatry. 2000 Mar;15(2):140-6. doi: 10.1016/s0924-9338(00)00219-4. PMID 10881212
- [Background] Le Foll B, Goldberg SR, Sokoloff P. Dopamine D3 receptor ligands for the treatment of tobacco dependence. Expert Opin Investig Drugs. 2007 Jan;16(1):45-57. doi: 10.1517/13543784.16.1.45. PMID 17155853
- [Background] Brody AL, Mandelkern MA, Olmstead RE, Scheibal D, Hahn E, Shiraga S, Zamora-Paja E, Farahi J, Saxena S, London ED, McCracken JT. Gene variants of brain dopamine pathways and smoking-induced dopamine release in the ventral caudate/nucleus accumbens. Arch Gen Psychiatry. 2006 Jul;63(7):808-16. doi: 10.1001/archpsyc.63.7.808. PMID 16818870
- [Background] Boileau I, Guttman M, Rusjan P, Adams JR, Houle S, Tong J, Hornykiewicz O, Furukawa Y, Wilson AA, Kapur S, Kish SJ. Decreased binding of the D3 dopamine receptor-preferring ligand [11C]-(+)-PHNO in drug-naive Parkinson's disease. Brain. 2009 May;132(Pt 5):1366-75. doi: 10.1093/brain/awn337. Epub 2009 Jan 19. PMID 19153147
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research